CLINICAL TRIAL: NCT05526625
Title: Comparison Of Ultrasound-Based Measures Of Inferior Vena Cava And Internal Jugular Vein For Prediction Of Hypotension During Induction Of General Anesthesia
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ismail Fathy Ahmed Mohammed, M.Sc, Cairo University
Other Study IDs: MD-13-2020
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Ultrasound Based IVC IJV

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasound-based measurements of IVC & IJV. — Ultrasound-based measurements of IVC & IJV.

SUMMARY:
Hypotension after induction of general anesthesia is a frequent event in routine practice. Even a short period of hypotension may lead to tissue hypoperfusion and predispose to postoperative complications. Intra-operative hypotension is associated with renal injury, ischemic stroke, myocardial injury and postoperative mortality in patients having non-cardiac surgery under general anesthesia. Underlying hypovolemia is an important and modifiable risk factor for hypotension after anesthetics administration. Ultrasonographic studies of the inferior vena cava (IVC) and the internal jugular vein (IJV) for evaluation of intravascular volume status and prediction of hypotension during induction of general anesthesia have been established.

The present study was designed to compare, on ultrasound-based measures, between inferior vena cava and internal jugular vein for prediction of prolonged hypotension during induction of general anesthesia. The study was conducted at Kasr Al-Ainy hospital, Cairo University in Patients undergoing elective non-cardiac surgery under general anesthesia.

DETAILED DESCRIPTION:
Upon arrival to the operating room, routine monitors in the form of pulse oximetry, electrocardiogarm and non-invasive blood pressure monitors were applied. Intravenous line was secured and routine premedications (ranitidine 50 mg and ondansetron 4 mg) were administered.

IVC evaluation was done for the patients in the supine position. The examination was performed after 5 minutes rest. A curved ultrasound transducer set to abdominal mode (1-5 MHz; Acuson x300; Siemens Healthcare, Seoul, Korea) was placed in the subcostal area to visualize the IVC in the paramedian long-axis view. The IVC was visualized using two-dimensional mode as it enters the right atrium; then, pulse wave doppler was used to differentiate the IVC from the aorta. Respiratory variations of the IVC diameter were evaluated using M-mode imaging at medium sweep speed 2 to 3 cm distal to the right atrium. The measures were obtained 3 times and their average was calculated. Maximum and minimum IVC diameters over a single respiratory cycle were used to calculate the collapsibility index as follows:

(dIVCmax- dIVCmin)/dIVCmax Collapsibility index was expressed as a percentage.

IJV measurements were obtained in the supine position using a linear ultrasound transducer (5 - 13 MHz; Acuson x300; Siemens Healthcare, Seoul, Korea). The probe was placed horizontally at the middle level of the thyroid cartilage. After obtaining a clear transverse view of the right IJV, the IJV area was measured. The measures were repeated after changing the patient's position to the 10° Trendelenburg position. The maximum area of the IJV in the supine and Trendelenburg positions was recorded and the rate of change in IJV area was calculated as follows:

IJV change rate with posture = (IJV area in Trendelenburg position - IJV area in supine position)/(IJV area in Trendelenburg position) All ultrasonographic measurements were performed by a single trained anesthesiologist.

IJV measurements were obtained in the supine position using a linear ultrasound transducer (5 - 13 MHz; Acuson x300; Siemens Healthcare, Seoul, Korea). The probe was placed horizontally at the middle level of the thyroid cartilage. After obtaining a clear transverse view of the right IJV, the IJV area was measured. The measures were repeated after changing the patient's position to the 10° Trendelenburg position. The maximum area of the IJV in the supine and Trendelenburg positions was recorded and the rate of change in IJV area was calculated as follows:

IJV change rate with posture = (IJV area in Trendelenburg position - IJV area in supine position)/(IJV area in Trendelenburg position) All ultrasonographic measurements were performed by a single trained anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 50 years old
* Any scheduled non-cardiac surgery under general anesthesia
* ASA I, II

Exclusion Criteria:

* Patients with major vascular disease
* Unstable angina
* Ejection fraction < 40 %
* Respiratory distress
* Increased intra-abdominal pressure.
* Diabetes mellitus
* Implanted pacemaker
* Patients on ACEI or ARB
* Anticipated difficult intubation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing elective non-cardiac surgery under general anesthesia in Kasr Al-Ainy hospital.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the accuracy of IVC and IJV variations in prediction of prolonged post-induction hypotension. | Intra-operative along the time of the study
  Comparison of the accuracy (area under receiver operating characteristic curves) of IVC and IJV variations in prediction of prolonged post-induction hypotension (defined as MBP < 80% of the baseline reading for 2 minutes or more).

SECONDARY OUTCOMES:
Incidence of prolonged post-induction hypotension. | Intra-operative along the time of the study
  Incidence of prolonged post-induction hypotension.
The accuracy of maximum diameter of IVC in predicting prolonged post-induction hypotension. | Intra-operative along the time of the study
  The accuracy of maximum diameter of IVC in predicting prolonged post-induction hypotension.
The accuracy of minimum diameter of IVC in predicting prolonged post-induction hypotension. | Intra-operative along the time of the study
  The accuracy of minimum diameter of IVC in predicting prolonged post-induction hypotension.
The accuracy of IVC collapsibility index in predicting prolonged post-induction hypotension. | Intra-operative along the time of the study
  The accuracy of IVC collapsibility index in predicting prolonged post-induction hypotension.
The accuracy of IJV area in supine position in predicting prolonged post-induction hypotension. | Intra-operative along the time of the study
  The accuracy of IJV area in supine position in predicting prolonged post-induction hypotension.
The accuracy of IJV area in Trendelenburg position in predicting prolonged post-induction hypotension. | Intra-operative along the time of the study
  The accuracy of IJV area in Trendelenburg position in predicting prolonged post-induction hypotension.
The accuracy of IJV change rate in predicting prolonged post-induction hypotension. | Intra-operative along the time of the study
  The accuracy of IJV change rate in predicting prolonged post-induction hypotension.
Incidence of severe post-induction hypotension. | Intra-operative along the time of the study
  Incidence of severe post-induction hypotension (defined as MBP < 60% of the baseline preoperative reading) until 15 minutes after anesthetics administration or until skin incision whichever is earlier.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al-ainy hospital, Cairo, Cairo Government, Egypt

IPD SHARING:
Plan to Share IPD: No